CLINICAL TRIAL: NCT01988324
Title: Androgen Receptor and Estrogen Receptor Imaging in Metastatic Breast Cancer Patients
Brief Title: AR and ER Imaging in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012.2708
Record Dates: First submitted 2013-11-01; First posted 2013-11-20 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

ARMS (1):
- FES/FDHT-PET (Experimental)
  Interventions: Other: FDHT-PET scan; Other: FES-PET scan; Other: CT-scan; Other: Bone scintigraphy; Other: Tumor biopsy

INTERVENTIONS:
Other: FDHT-PET scan
Other: FES-PET scan
Other: CT-scan
Other: Bone scintigraphy
Other: Tumor biopsy

SUMMARY:
Knowledge of breast cancer estrogen receptor (ER) expression is of major importance in treatment-decision making. Patients with ER-positive tumors can be treated with anti-oestrogen therapy, which has relatively few side effects compared to chemotherapy. Whole-body tumor ER-expression can be visualized by 18F-fluoroestradiol PET imaging (FES-PET). In addition to ER, the androgen receptor (AR) is a potential new target in breast cancer. PET imaging with 18F-fluorodihydrotestosterone (18F-FDHT) may allow visualization of tumor AR-expression. In the current study we will perform FES-PET and FDHT-PET in metastatic breast cancer patients and evaluate the concordance with concurrent biopsies. Molecular imaging of tumor AR- and ER-expression may well be of value for future treatment decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic breast cancer, with at least one known metastasis outside of the liver
2. Presence of a lesion that is safely accessible for tumor biopsy (may be liver lesion)
3. Postmenopausal status defined as one of the following:

   * age ≥60 years
   * previous bilateral oophorectomy
   * age <60 years and amenorrhea for >12 months in the absence of interfering hormonal therapies (such as LH-RH agonists and ER-antagonists)
   * patients age <60 years using an ER-antagonist should have amenorrhea for > 12 months and FSH >24 U/L and LH >14 U/L e. patient age <60 years using LH-RH agonists should continue LH-RH-agonists until after the PET procedures
4. Initially ER-positive tumor histology.
5. ECOG performance status 0-2.
6. Signed written informed consent
7. Able to comply with the protocol

Exclusion Criteria:

1. Use of estrogen receptor ligands, including tamoxifen, fulvestrant or estrogens, or androgen receptor ligands, during the 6 weeks before entry into the study
2. Life-expectancy ≤ 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity/ specificity | within two months
  The concordance between PET (with 18F-FDHT and 18F-FES), and immunohistochemistry (for AR and ER) on concurrent (within 8 weeks) tumor biopsy will be evaluated.

SECONDARY OUTCOMES:
Accuracy | within six weeks
  The number of lesions detected on PET imaging compared to CT-scan and bone scintigraphy.
Inter- and intra-patient variation | within six weeks
  Inter- and intra-patient variation in tumor FDHT and FES-uptake will be calculated.
Inter-observer variation | approximately two months
  Inter-observer variation in FES PET and FDHT PET results in two independent observers.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - VU Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen

REFERENCES:
- [Derived] Mammatas LH, Venema CM, Schroder CP, de Vet HCW, van Kruchten M, Glaudemans AWJM, Yaqub MM, Verheul HMW, Boven E, van der Vegt B, de Vries EFJ, de Vries EGE, Hoekstra OS, Hospers GAP, der Houven van Oordt CWM. Visual and quantitative evaluation of [18F]FES and [18F]FDHT PET in patients with metastatic breast cancer: an interobserver variability study. EJNMMI Res. 2020 Apr 19;10(1):40. doi: 10.1186/s13550-020-00627-z. PMID 32307594